CLINICAL TRIAL: NCT05984433
Title: Auricular Acupuncture As Part Of A Multimodal Analgesic Regimen For Reduction Of Opioid Analgesic Use After Surgery To Repair Lower Leg Fractures- A Randomized Controlled Trial
Brief Title: Auricular Acupuncture as Part of Multimodal Analgesia After Lower Leg Fracture
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Baylor College of Medicine (Other)
Responsible Party: Principal Investigator, Jaime Ortiz, Professor of Anesthesiology, Baylor College of Medicine
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: H-53820
Record Dates: First submitted 2023-07-26; First posted 2023-08-09 (Actual); Last update posted 2025-01-14 (Actual); Status verified 2025-01

CONDITIONS: Pain, Postoperative; Fracture, Ankle; Pilon Fracture of Tibia; Foot Fracture
MeSH Terms: conditions — Pain, Postoperative; Ankle Fractures | interventions — Acupuncture, Ear

STUDY DESIGN:
Intervention Model Description: Randomized controlled trial. Group 1 - acupuncture Group 2 - no acupuncture 70 patients per group
Who Masked: Participant, Outcomes Assessor
Masking Description: The patient will be under sedation during procedure, so will not be aware of whether or not they received acupuncture treatment.
  Anesthesia team in the operating room will be aware of treatment. PACU team and outcomes assessor will not be aware of group assignment
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

ARMS (2):
- Electroauricular acupuncture (Experimental): Immediately after Level 2 sedation is achieved, an enhanced auricular trauma protocol (ATP) will be administered on the ear ipsilateral to the operative side at 8 ear points (Hypothalamus, Amygdala, Hippocampus, Prefrontal Cortex, Point Zero, Shen Men, Insula, Vagus) as described by Cheng (2022). The original ATP was described by Helms (2011). Seirin L 0.2 x 30 mm needles will be placed at Hypothalamus and Shen Men points. Seirin J 0.18 x 15 mm needles will be placed at Amygdala, Hippocampus, Prefrontal Cortex, Point Zero, Vagus, and Insula points. Electrostimulation using an ITO ES 130 microstimulator at 30 HZ with Level 4 intensity, will be applied with the positive lead (red) on Hypothalamus and negative lead (black) at Shen Men for 60 minutes. All needles will be removed 1 hour after insertion.
  Interventions: Device: Auricular acupuncture
- No acupuncture (No Intervention): No acupuncture treatment given

INTERVENTIONS:
Device: Auricular acupuncture — Electro auricular acupuncture
  Arms: Electroauricular acupuncture

SUMMARY:
The purpose is to find out if incorporation of an intraoperative electro auricular acupuncture protocol when added to a standard multimodal analgesic regimen for patients undergoing surgery to repair lower leg fracture under spinal anesthesia will help reduce postoperative opioid use.

ELIGIBILITY:
Inclusion Criteria:

1. Patient ages 18-64
2. American Society of Anesthesiology Physical Status I, II or III
3. Inpatients scheduled to undergo ankle ORIF at Harris Health System Ben Taub Hospital

Exclusion Criteria:

1. Renal dysfunction (Serum Cr > 1.2) - excluded due to potential altered metabolism of anesthetic and perioperative medications
2. Allergy to any of the standard anesthetic agents
3. Patient inability to properly communicate with investigators (language barrier, dementia, delirium, psychiatric disorder)
4. Patient or surgeon refusal

Ages: 18 Years to 64 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 140 (Estimated)
Dates: Start 2024-10-09 (Actual); Primary Completion 2026-12 (Estimated); Study Completion 2026-12 (Estimated)

PRIMARY OUTCOMES:
Total opioid analgesic use for 14 days after surgery | 14 days
  Total opioid given in hospital and taken at home, converted to oral morphine equivalents

SECONDARY OUTCOMES:
Pain scores | 14 days
  Pain scores (1-10) in PACU and at the 7 and 14 day mark post surgery
Incidence of side effects associated with opioid use | 14 days
  PONV, pruritus, headache, constipation, urinary retention, fatigue, difficulty with concentration, drowsiness, lightheadedness, dry mouth

CONTACTS AND LOCATIONS:
Locations (1):
- Ben Taub Hospital, Houston, Texas, United States

IPD SHARING:
Plan to Share IPD: No